CLINICAL TRIAL: NCT04585295
Title: The Effects of Pre-Loaded Betaine Supplementation on Thermoregulation and Exercise Metabolism in the Heat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: NOW Foods (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Principal Investigator, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Betaine
Record Dates: First submitted 2019-07-08; First posted 2020-10-14 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Betaine; NOW Foods BCAA Big 6; Placebo
MeSH Terms: interventions — Betaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Betaine (Experimental): Aim 1: To evaluate the impact of preloaded betaine supplementation on fluid compartments in male athletes aged 18-45 years old.
  Aim 2: To determine the degree to which preloading with betaine impacts heat tolerance relative to placebo in male athletes aged 18-45 years old.
  Aim 3: To determine the degree to which preloading with betaine impacts exercise metabolism and performance in the heat relative to placebo in male athletes aged 18-45 years old.
  Interventions: Dietary Supplement: Betaine; Dietary Supplement: BCAA Big 6; Dietary Supplement: Placebo
- Placebo (Experimental): Aim 1: To evaluate the impact of preloaded betaine supplementation on fluid compartments in male athletes aged 18-45 years old.
  Aim 2: To determine the degree to which preloading with betaine impacts heat tolerance relative to placebo in male athletes aged 18-45 years old.
  Aim 3: To determine the degree to which preloading with betaine impacts exercise metabolism and performance in the heat relative to placebo in male athletes aged 18-45 years old.
  Interventions: Dietary Supplement: Betaine; Dietary Supplement: BCAA Big 6; Dietary Supplement: Placebo
- NOW Foods Big 6 (Experimental): Aim 1: To evaluate the impact of preloaded betaine supplementation on fluid compartments in male athletes aged 18-45 years old.
  Aim 2: To determine the degree to which preloading with betaine impacts heat tolerance relative to placebo in male athletes aged 18-45 years old.
  Aim 3: To determine the degree to which preloading with betaine impacts exercise metabolism and performance in the heat relative to placebo in male athletes aged 18-45 years old.
  Interventions: Dietary Supplement: Betaine; Dietary Supplement: BCAA Big 6; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Betaine — 50 mg/kg Betaine consumed twice daily for 7 days.
  Other Names: Trimethylglycine
Dietary Supplement: BCAA Big 6 — 1 level scoop (~18 g) of NOW Foods BCAA Big 6, consumed once per day for 7 days.
Dietary Supplement: Placebo — 50 mg/kg Placebo consumed twice daily for 7 days.

SUMMARY:
This will be a double blind, placebo-controlled, randomized, counterbalanced, crossover study designed to assess the impact of preloaded betaine supplementation on thermoregulation and exercise metabolism in the heat. The study, outlined in Figure 7 and described in detail below, will consist of seven total visits to the Institute of Sports Science and Medicine (ISSM) or Sandels laboratories at Florida State University, two of which will be experimental visits. On the first visit, participants will be informed as to the details of the study before giving their oral and written informed consent (Appendix A). Thereafter, anthropometrics will be measured and participants will complete an incremental exercise test on an electronically-braked cycle ergometer to volitional exhaustion to determine peak oxygen consumption (VO2 peak). Days 1-6 participants will consume a full dosage of supplementation, whereas day 0 and 7 participants will consume half a dose of the supplement, with the last dosage being consumed 60 minutes prior to experimental visits, days 7 and 21. On days 2 and 4, familiarization trials will be completed to standardize training loads and to reduce any potential learning effect. These visits will be implemented in the heat. On day 7, participants will complete the first experimental trial described in detail below. Afterwards, participants will enter a seven day washout period 167 before crossing over to the second supplemental condition on day 14. On days 16 and 18, participants will undergo the same familiarization trials as they did on days 2 and 4. On day 21, participants will complete their second experimental trial. Each experimental trial will be separated by 14 days. This study will be approved by the Florida State University Insitutional Review Board (Appendix B).

DETAILED DESCRIPTION:
Initial Visit Participants will be asked to come into the ISSM in the morning, following an overnight fast (7-9 hr) having abstained from caffeine for the previous 12 hours, and having abstained from alcohol and exercise for the previous 24 hr. Participants will be asked to consume 6 ml·kg-1 water 60 minutes prior to arrival. Following the signing of the informed consent document, participants will be asked to change into athletic clothing. Thereafter, with shoes removed, participants' height will be assessed to the nearest cm via a wall-mounted scale (Seca, Hamburg, Germany). Participants will be weighed to the nearest 0.1 kg via an automated scale (Detecto® 750, Webb City, MO). Body composition will then be assessed via Bod Pod (Cosmed, Chicago, IL). Participants will be asked to rest quietly in a supine position for 5 minutes, before blood pressure will be measured via auscultation and sphygmomanometry (Grainger, Lake Forest, Illinois). While still in a supine position, fluid compartments will be measured via bioelectric impedance spectroscopy (BIS) (ImpediMed SFB7, ImpediMed Limited, Australia).

Following these baseline measurements, participants will be asked to wear a heart rate monitor then complete a self-determined 5-min warm-up on an electronically-braked cycle ergometer (Velotron, SRAM, Spearfish, SD). Immediately after the warm-up, participants will be fitted with a metabolic mask (TrueOne 2400 Metabolic Cart, ParvoMedics, Sandy, Utah) then commence an incremental exercise test to exhaustion. The incremental test will consist of 3-min stages in which the resistance will begin at a relative intensity of 2 W·kg-1 and increase in 25 W increments until RER is greater than 1.0. At this point, the test will switch to 1-min stages with resistance increasing in 10 W increments until volitional exhaustion. A similar protocol is described elsewhere 223.

Afterwards, participants will be provided with their blinded supplement and instructed to consume 50 mg·kg-1 twice daily (~12 hr apart) with 6 ml·kg-1 water each time, for 7 days.

Familiarization Trials The familiarization trials will occur the first week of supplementation on days 2 and 4, and the second week of supplementation on days 16 and 18. On familiarization days, participants will be asked to arrive at the Sandels building in the morning in a euhydrated state, having consumed 6 ml·kg-1 water 60 minutes prior to arrival. Additionally, participants will be asked to arrive following an overnight fast (7-9 hr) having abstained from caffeine for the previous 12 hours, and having abstained from alcohol and exercise for the previous 24 hr. Upon arrival, the participant will be fitted with a heart rate monitor (Polar® FT4M, Sempele, Finland). Participants will enter the chamber (33° C, 35% RH), be fitted with a metabolic mask (TrueOne 2400 Metabolic Cart, ParvoMedics, Sandy, Utah) and cycle for 30 min at 70% VO2 peak. After a 5 min active recovery period, self-paced pedaling against 50 W, participants will perform four 12 s maximal effort sprints against 5.5% of their body mass, followed by one 30 s maximal effort sprint against 5.5% of their body mass. Participants will perform 2.5 min active recovery (self-paced pedaling against 50 W) between sprints. Participants will then exit the chamber and be allowed to drink ad libitum in a resting position.

Experimental Trials This section provides an overview of the experimental trials, with greater detail provided in the appropriate sections below.

The experimental trials will occur after the first week of supplementation on day 7, and the second week of supplementation on day 21. The participants will be asked to ingest a CorTemp Sensor (HQInc, Palmetto, FL) 10-12 hr before arrival. Participants will be asked to arrive at the Sandels building in the morning in a euhydrated state, having consumed 6 ml·kg-1 water 60 minutes prior to arrival. Additionally, participants will be asked to arrive following an overnight fast (7-9 hr) having abstained from caffeine for the previous 12 hours, and having abstained from alcohol and exercise for the previous 24 hr. Participants will be asked to provide a urine sample to confirm hydration status. A urine specific gravity (USG) measurement of >1.020 will be considered dehydrated, whereas a USG measurement of <1.020 will be considered euhydrated 124-126. If the participant is considered dehydrated upon arrival, they will be provided with 6 mL·kg-1 water and the experimental trial will be pushed back another 30 minutes. Additionally, hydration status will be measured via changes in pre- to post-exercise body mass. Participants, in a private room, will be asked to towel dry and provide a nude body weight while resting pre-exercise, and again after the 60 min bout of exercise. Prior to exercise, participants will be asked to rest quietly in a supine position for 5 minutes, before blood pressure will be measured via auscultation and sphygmomanometry (Grainger, Lake Forest, Illinois). While still in a supine position, fluid compartments will be measured via bioelectric impedance spectroscopy (BIS) (ImpediMed SFB7, ImpediMed Limited, Australia).

Participants will then be fitted with iButtons (iButton DS1921G-F5, Maxim Integrated, San Jose, CA, USA) to estimate whole body skin temperature from 7 standardized locations on the body. Specifically, the investigators will use the abdomen (site A), inferior angle of the left scapula (site B), left posterior forearm (site C), dorsal side of the left hand (site D), left anterior thigh (site E), posterior side of the lower leg (site F), and left mid-foot (site G) 224. Then, participants will be seated in an upright position and fitted with a heart rate monitor (Polar® FT4M, Sempele, Finland) and metabolic mask (TrueOne 2400 Metabolic Cart, ParvoMedics, Sandy, Utah). Baseline measures of core temperature, skin temperature, heart rate, gas exchange, and blood will be sampled at this time.

Following baseline measurements, participants will enter the chamber (33° C, 35% RH) and complete a workload corresponding to 70% VO2 peak for 60 min. Immediately following the steady state exercise bout, participants will have a 5 min rest period to collect a blood sample and nude body weight. Afterwards, participants will perform four 12 s maximal effort sprints against 5.5% of their body mass, followed by one 30 s maximal effort sprint against 5.5% of their body mass. Participants will perform 2.5 min active recovery (self-paced pedaling against 50 W) between sprints. Participants will then exit the chamber and be allowed to drink ad libitum in a resting position.

Environmental Chamber Ambient Temperature Ambient temperature and humidity will be controlled via the environmental chamber and will be secondarily confirmed (Vantage Vue Weather Station, Davis Instruments, Hayward, California) in 10 min increments throughout experimental visits.

Standardization of Diet and Training Prior to each familiarization and experimental visit, participants will be asked to maintain consistent dietary and exercise habits for 2 days. Additionally, for both days leading up to experimental trials, participants will be asked to exactly replicate their dietary intake from week to week. To ensure compliance, participants will be asked to complete a 48-hr dietary intake form (Appendix C) and a 48-hr exercise log (Appendix D) for the days preceding the experimental trial. Finally, participants will be asked to abstain from caffeine for the previous 12 hours, and abstain from alcohol and exercise for the previous 24 hr.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male
2. Age: 18-45 yr
3. Trained male cyclists: ≥ 3 yr cycling experience
4. Participants' VO2 peak > 50.0 ml·kg·min-1

Exclusion Criteria:

1. Sex: female
2. Age: < 18 yr or > 45 yr
3. Cigarette smoking: current cigarette smoker or those who quit within the previous 6 months
4. Participants' VO2 peak < 50.0 ml·kg·min-1
5. Participants consuming supplements known to impact hydration status and exercise performance
6. Participants known to have sickle cell trait or disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Fluid Compartment Volumes (Bioelectrical Impedance Spectrocopy) | pre and post 7 days of supplementation
  Intracellular fluid volume (L), extracellular fluid volume (L), plasma volume (L), total body water (L)
Thermoregulation (core temperature pills, skin temperature sensors) | pre and post 7 days of supplementation & minutes 0, 15, 30, 45, 60, 75, and 90 during the experimental visit
  Core temperature (Degrees C), skin temperature (Degrees C)
Thermoregulation (enzyme linked immunoassays) | 7 days of supplementation & minutes 0, 30, 60, and 90 during the experimental visit
  serum expression of heat shock protein 72 and plasma lipopolysaccharide concentrations
Thermoregulation (thermal sensation scale) | minutes 0, 15, 30, 45, 60, 75, and 90 during the experimental visit
  Subjective self-reported assessment of perceived thermal sensation (arbitrary units)

SECONDARY OUTCOMES:
Exercise Metabolism and Performance (heart rate) | minutes 0, 15, 30, 45, 60, 75, and 90 during the experimental visit
  heart rate (beats per minute)
Exercise Metabolism and Performance (Oxygen Consumption) | minutes 0-5, 25-30, and 55-60 during the experimental visit
  volume of oxygen consumption (L), volume of carbon dioxide production (L)

CONTACTS AND LOCATIONS:
Overall Officials: Miachael Ormsbee, PhD, Study Director — Florida State University
Locations (1):
- Institute of Sport Sciences and Medicine at Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No